CLINICAL TRIAL: NCT02217332
Title: Safety and Preliminary Efficacy of Dexpramipexole in Patients With Chronic Sinusitis With Nasal Polyps and Eosinophilia (CSNP-E)
Brief Title: Study of Dexpramipexole Chronic Sinusitis With Nasal Polyps and Eosinophilia
Acronym: CS201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNS-76704-CS201
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Chronic Sinusitis With Nasal Polyps and Eosinophilia
Keywords: Sinusitis; Rhinosinusitis; CRS; CRSwNP; CSNP-E; Nasal polyps; Nasal polyposis; Eosinophilia; Asthma
MeSH Terms: conditions — Eosinophilia; Sinusitis; Rhinosinusitis; Nasal Polyps; Asthma | interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexpramipexole (Experimental): dexpramipexole 150 mg BID
  Interventions: Drug: dexpramipexole

INTERVENTIONS:
Drug: dexpramipexole — Dexpramipexole capsule-shaped film-coated tablets at the dose strength of 150 mg administered orally as 1 tablet twice daily (300 mg/day)
  Other Names: KNS-760704; BIIB050; RPPX

SUMMARY:
Phase 2, open-label, multi-center study to evaluate the clinical effects of oral administration of dexpramipexole for 6 months in subjects with chronic sinusitis with nasal polyps and eosinophilia.

DETAILED DESCRIPTION:
This open-labelled study will evaluate the safety and preliminary efficacy of dexpramipexole for reducing the number of eosinophils in the peripheral blood and in improving nasal polyp score when administered to 20 subjects with chronic sinusitis with nasal polyps and eosinophilia.

Subjects will received dexpramipexole for up to 6 months and will have safety tests performed monthly and will have efficacy evaluations performed at month 1, month 3, and month 6 after beginning study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 or <70 years of age
* Willing to practice effective contraception during the study and be willing and able to continue contraception for 1 month (females) or 3 months (males) after the last dose of study treatment
* Confirmed diagnosis of chronic sinusitis with nasal polyps
* Documented history of nasal eosinophilia
* Documented peripheral absolute eosinophil count >300 cells/μL
* Bilateral total polyp score of >4
* Sino-nasal outcome test (SNOT-22) score of >7
* Using an intranasal corticosteroid spray or irrigation (< 1000 μg/day beclomethasone or equivalent)

Exclusion Criteria:

* Acute sinusitis, concurrent nasal infection, or subjects who have had a nasal or upper respiratory tract infection within 2 weeks prior to baseline
* CT scan suggestive of allergic fungal rhinosinusitis
* Nasal septal deviation that would occlude at least one nostril
* Nasal surgery (including polypectomy) within 6 months prior to baseline
* History of more than 5 sinonasal surgeries requiring general anesthesia
* History of more than 2 sinonasal surgeries that changed the lateral wall of the nose
* History of cystic fibrosis, primary ciliary's dysfunction or Kartagener's syndrome
* History of diagnosis with a parasitic infection
* Hospitalization or emergency treatment for the treatment of asthma two or more times in the 12 months prior to baseline
* Hospitalization for an acute asthmatic attack within 4 weeks prior to baseline
* Forced expiratory volume (FEV1) of <60% of predicted normal range
* Treatment with a systemic corticosteroid or intra-polyp corticosteroid within 8 weeks prior to baseline or anticipated need for systemic corticosteroids during the study treatment period
* Utilization of rescue oral corticosteroids for asthma or chronic sinusitis exacerbation more than one time within the past 1 year
* Treatment with an investigational drug in the previous 30 days or 5-half-lives, whichever is longer
* Treatment with a monoclonal antibody therapy including omalizumab (Xolair®), within 5-half-lives
* Treatment with zileuton (Zyflo®) within 4 weeks of baseline
* Treatment with pramipexole (Mirapex®) within 4 weeks of baseline
* History of malignancy, including solid tumors and hematologic malignancies (except basal cell and squamous cell cancers of the skin that have been completely excised and cured)
* History of human immunodeficiency virus (HIV) or hepatitis B or C
* History of unstable or severe cardiac, hepatic, or renal disease, or other medically significant illness
* Medical or other condition likely to interfere with subject's ability to undergo study procedures, adhere to visit schedule or comply with study requirements
* Absolute neutrophil count <2000 cells/μL at screening, or any documented history of neutropenia
* Total IgE >1500 IU/ml at any visit prior to baseline
* Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) of ≤80 mg/dL at screening (estimation of creatinine clearance using the MDRD formula)
* History of long QT syndrome or arrhythmia
* Prolongation of QT/QTc interval (e.g., repeated demonstration of a QT/QTc interval >450 ms) at screening or pre-dose on day 1
* Clinically important abnormalities in resting ECG that may interfere with the interpretation of QTc interval changes at screening or pre-dose on day 1, including any of the following:

  * PR interval >210 ms;
  * QRS >110 ms;
  * Heart rate <45 bpm or >100 bpm (average of 3 assessments).
* Pregnant women or women breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-14 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - ENT Associates of South Florida, Boca Raton, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Wake Research Associates, Raleigh, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During a screening period of between 14 and 21 days, subjects were monitored symptoms of sinusitis and asthma. Subject who failed to meet the eligibility criteria during the screening period were disqualified.
Period: Overall Study
Arm/Group | Dexpramipexole
Started | 20 (Safety Population)
Completed | 13 (Subjects who continued to optional open-label treatment)
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Dose interruption >1 month | 1
Not completed — Protocol Violation (eligibility) | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (9.78)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 14
  50 to 65 years | 5
  > 65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
CSNP-E Symptoms [Count of Participants; unit: Participants]
  Anterior and/or posterior mucopurulent drainage | 20
  Sinonasal obstruction/congestion | 20
  Decreased sense of smell (anosmia) | 20
Duration of Symptoms (months) [Mean (Standard Deviation); unit: months] | 112.4 (138.13)
Duration of symptoms [Count of Participants; unit: Participants]
  ≤ 1 year | 3
  > 1 year to ≤ 5 years | 6
  > 5 years to ≤ 10 years | 6
  > 10 years | 5

OUTCOME MEASURES:

1. Primary Outcome: Ratio to Baseline in Peripheral Blood Eosinophil Counts After 6 Months of Treatment
Description: Change in peripheral blood eosinophil (measured in cells/μL) from baseline to month 6 is presented as ratio to baseline.
Time Frame: Baseline and Month 6
Population: All subjects who had a Month 3 evaluation (on study drug Day 77 or later) for TPS and peripheral blood eosinophil count. Last observation carried forward (LOCF) was used to replace missing data due to drop out. Only Month 3 data or later (assessment date Day 77 or later and within 7 days of last dose) were used.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio to baseline
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 16
ratio to baseline | 0.06 [0.023 to 0.154]
Statistical Analysis 1: Comparison: Dexpramipexole; Null hypothesis is the ratio of Month 6 to Baseline within the dexpramipexole group equals '1'; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired t-test comparing baseline to month 6 on log scale within the dexpramipexole treatment group

2. Primary Outcome: Change From Baseline in Total Polyp Score (TPS) After 6 Months of Treatment
Description: The change in Nasal Polyp Score (NPS) score after 6 months of treatment is presented. A blinded Central Endoscopy Rater determined the NPS for each nare on a scale of 0 to 4, and the bilateral NPS scores were added to generate the Total Polyp Score (TPS) on a scale of 0 to 8. A lower TPS corresponds to a lower polyp burden.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 15
units on a scale | 0.07 (1.751)
Statistical Analysis 1: Comparison: Dexpramipexole; Test type: Superiority; p = 0.885, t-test, 2 sided — Month 6/LOCF was used for the analysis of change from Baseline to Month 6 within the dexpramipexole group

3. Secondary Outcome: Number of Subjects With Potentially Clinically Significant Values in Clinical Laboratory Evaluations
Description: Summary of subjects from the safety population who experienced potentially clinically significant values in hand serum chemistry results
Time Frame: 6 months
Population: The safety population included all subjects who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 20
Participants
  LOW: Albumin <= 25 g/L | 0
  HIGH: Alanine aminotransferase (ALT) >= 1.5 x ULN | 1
  HIGH: Aspartate aminotransferase (AST) >= 1.5 x ULN | 0
  HIGH: Total bilirubin >= 1.5 x ULN | 0
  HIGH: Glucose>= 9.7 mmol/L | 1
  LOW: Glucose <= 2.2 mmol/L | 1
  HIGH: Eosinophils > 1.6 x 10(9)/L | 1
  HIGH: Hematocrit - Females >=54%: number analyzed (Participants) | 8
  HIGH: Hematocrit - Females >=54% | 0
  LOW: Hematocrit - Females <= 32%: number analyzed (Participants) | 8
  LOW: Hematocrit - Females <= 32% | 2
  HIGH: Hemoglobin - Females >=175g/L: number analyzed (Participants) | 8
  HIGH: Hemoglobin - Females >=175g/L | 0
  LOW: Hemoglobin - Females <= 95g/L: number analyzed (Participants) | 8
  LOW: Hemoglobin - Females <= 95g/L | 2
  HIGH: Lymphocytes > 12 x 10(9)/L | 0
  LOW: Lymphocytes < 0.8 x 10(9)/L | 2
  LOW: Neutrophils < 1.5 x 10(9)/L | 0

4. Secondary Outcome: Number of Subjects With Potentially Clinically Significant Values in Vital Signs and Weight
Description: Summary of subjects from the safety population who experienced potentially clinically significant values or changes in vital signs or weight
Time Frame: 6 months
Population: The safety population included all subjects who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 20
Participants
  Systolic Blood Pressure: >180 mmHg | 0
  Systolic Blood Pressure: increase from pre-dosing of more than 40 mmHg | 0
  Systolic Blood Pressure: <90 mmHg | 0
  Systolic Blood Pressure: decrease from pre-dosing of more than 30 mmHg | 0
  Diastolic Blood Pressure: >105 mmHg | 0
  Diastolic Blood Pressure: increase from pre-dosing of more than 30 mmHg | 0
  Diastolic Blood Pressure: <50 mmHg | 0
  Diastolic Blood Pressure: decrease from pre-dosing of more than 20 mmHg | 0
  Heart Rate: >120 beats per minute | 0
  Heart Rate: increase from pre-dosing of more than 20 beats per minute | 1
  Heart Rate: <50 beats per minute | 0
  Heart Rate: decrease from pre-dosing of more than 20 beats per minute | 0
  Temperature: >38ºC and an increase from pre-dosing of at least 1ºC | 0
  Body Weight: >7% increase from baseline value | 0
  Body Weight: <=7% decrease from baseline value | 0

5. Secondary Outcome: Number of Subjects With Potentially Significant Values in Electrocardiogram Parameters
Description: Summary of subjects from the safety population who experienced potentially significant values in electrocardiogram parameters
Time Frame: 6 months
Population: The safety population included all subjects who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 20
Participants
  QTcF: >450 msec | 2
  QTcF: >480 msec | 0
  QTcF: > 450 msec and ≤ 450 msec at baseline | 1
  QTcF: > 480 msec and ≤ 480 msec at baseline | 0
  QTcF: > 450 msec and change from baseline > 30 msec | 0
  QTcF: > 480 msec and change from baseline > 30 msec | 0
  QTcF change from baseline: >30 msec | 1
  QTcF change from baseline: >60 msec | 0
  Rhythm abnormalities: Sinus rhythm | 17
  Rhythm abnormalities: Sinus bradycardia | 3
  Rhythm abnormalities: Premature atrial complexes, conducted or non-conducted sinus rhythm | 1
  ST-T abnormalities: Nonspecific T wave abnormality | 3
  ST-T abnormalities: Early repolarization | 1
  ST-T abnormalities: Early repolarization, considered normal variant | 1
  ST-T abnormalities: Nonspecific ST deviation | 1
  ST-T abnormalities: Nonspecific ST deviation, prolonged QTcF interval | 1
  ST-T abnormalities: Nonspecific T wave abnormality, prolonged QTcF interval | 1
  ST-T abnormalities: Prolonged QTcF interval | 1
  Conduction abnormality: First degree AV block | 2
  Conduction abnormality: Complete right bundle branch block | 1
  Conduction abnormality: Complete right bundle branch block first degree AV block | 1

6. Secondary Outcome: Ratio to Baseline in Peripheral Blood Eosinophil Counts After 3 Months of Treatment
Description: Change in peripheral blood eosinophil (measured in cells/μL) from baseline to month 3 is presented as ratio to baseline.
Time Frame: Baseline and Month 3
Population: All subjects who had a Month 3 evaluation (on study drug Day 77 or later) for total eosinophil count
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 16
ratio | 0.05 [0.019 to 0.142]
Statistical Analysis 1: Comparison: Dexpramipexole; Null hypothesis is the ratio of Month 3 to Baseline within the dexpramipexole group equals '1'; Test type: Superiority; p < .001, t-test, 2 sided; Paired t-test comparing baseline to month 3 on log scale within the dexpramipexole treatment group

7. Secondary Outcome: Change From Baseline in TPS After 3 Months of Treatment
Description: The change in Nasal Polyp Score (NPS) score after 3 months of treatment is presented. A blinded Central Endoscopy Rater determined the NPS for each nare on a scale of 0 to 4, and the bilateral NPS scores were added to generate the Total Polyp Score (TPS) on a scale of 0 to 8. A lower TPS corresponds to a lower polyp burden.
Time Frame: Baseline and Month 3
Population: All subjects who had a Month 3 evaluation (on study drug Day 77 or later) for total eosinophil count and total polyp score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 16
units on a scale | 0.0 (1.414)
Statistical Analysis 1: Comparison: Dexpramipexole; Test type: Superiority; p = 1.0, t-test, 2 sided — Month 3/LOCF was used for the analysis of change from Baseline to Month 3 within the dexpramipexole group; Paired t-test comparing baseline to month 3 within the dexpramipexole treatment group

8. Other Pre Specified Outcome: Ratio to Baseline in Polyp Tissue Eosinophil Count After 6 Months of Treatment
Description: Change in polyp tissue eosinophil count measured as eosinophils/hpf (high powered field) from baseline to month 6 is presented as ratio to baseline.
Time Frame: Baseline and Month 6
Population: All subjects who had a Month 3 evaluation (on study drug Day 77 or later) for TPS and peripheral blood eosinophil count (Efficacy Population). Additionally, subjects with <5 eos/hpf at screening or baseline visit are not included in this analysis.
Measure: Geometric Mean (68% Confidence Interval); unit: ratio to baseline
Arm/Group | Dexpramipexole
Number analyzed (Participants) | 12
ratio to baseline | 0.03 [0.02 to .06]
Statistical Analysis 1: Comparison: Dexpramipexole; Null hypothesis is the ratio of Month 6 to Baseline within the dexpramipexole group equals '1'; 68% confidence interval is equal to plus/minus 1 standard error; Test type: Superiority; p = 0.001, Wilcoxon Signed Rank Test (paired); log scale

ADVERSE EVENTS:
Time Frame: 6 months on treatment
Arm/Group | Dexpramipexole
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexpramipexole (N=20)
biliary dyskinesia (Metabolism and nutrition disorders) | 1 (1) — The investigator and the sponsor both assessed the SAE of cholecystitis as not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexpramipexole (N=20)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Xerosis (General disorders) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4)
Onychomycosis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 8 (12)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intranasal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other